CLINICAL TRIAL: NCT03669276
Title: Effect of Gonadotropin Types and Indications on Homologous Intrauterine Insemination Success: A Study From 1251 Cycles and a Review of the Literature
Brief Title: Effect of Gonadotropin Types and Indications on Homologous Intrauterine Insemination Success
Acronym: GONADOTROP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0046
Record Dates: First submitted 2018-08-27; First posted 2018-09-13 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators took the opportunity of having a large sample of IUI cycles in a single centre to try to analyse the effect of stimulation protocols and of the infertility origin on the results, taking in account the main confounding variables (female age, IUI attempt rank, and sperm quality) on the clinical outcome.

All couples had undergone a standard infertility evaluation, which included medical history, physical examination, and assessment of tubal patency by either hysterosalpingography or laparoscopy and hormonal analysis on cycle day 3. A transvaginal ultrasound scan was performed on the second day of the cycle. On the same day, ovarian stimulation was carried out with recombinant FSH (follitropinrFSH; Gonal-F, MerckSerono, France, orfollitropin;Puregon, MSD, France), urinary FSH (urofollitropin, Fostimon, France), orhMG (menotropin, Menopur, France) atastarting dose of 75 IU/day from the second day of the cycle.

The main clinical outcome measures were clinical pregnancy and live-birth rates per cycle. Clinical pregnancy was defined as the evidence of pregnancy by ultrasound examination of the gestational sac at weeks 5-7.

DETAILED DESCRIPTION:
Many studies have evaluated the predictive factors of IUI clinical outcomes, including the female's age, the infertility duration, the rank of the attempt, and the sperm parameters [10-16]. However, few studies have compared the pregnancy rates based on the used COS or on the infertility type.

In this study the investigators took the opportunity of having a large sample of IUI cycles in a single centre to try to analyse the effect of stimulation protocols and of the infertility origin on the results, taking in account the main confounding variables (female age, IUI attempt rank, and sperm quality) on the clinical outcome.

All couples had undergone a standard infertility evaluation, which included medical history, physical examination, and assessment of tubal patency by either hysterosalpingography or laparoscopy and hormonal analysis on cycle day 3. A transvaginal ultrasound scan was performed on the second day of the cycle. On the same day, ovarian stimulation was carried out with recombinant FSH (follitropinrFSH; Gonal-F, MerckSerono, France, orfollitropin;Puregon, MSD, France), urinary FSH (urofollitropin, Fostimon, France), orhMG (menotropin, Menopur, France) atastarting dose of 75 IU/day from the second day of the cycle.

The main clinical outcome measures were clinical pregnancy and live-birth rates per cycle. Clinical pregnancy was defined as the evidence of pregnancy by ultrasound examination of the gestational sac at weeks 5-7.

ELIGIBILITY:
Inclusion Criteria:

* women with a failure to conceive after, ≥12 months of unprotected and regular intercourse,
* aged 20-44 years
* with normal ovulation reserve (basal follicle- stimulating hormone (FSH) level < 10 IU/l and estradiol (E2) level < 30ng/mL);
* theirpartnershadtohaveatotal motile sperm (TMS) count of>1×106.

Exclusion Criteria:

* TMS ≤1×106;
* sperm donation;
* seropositivity for human immunodeficiency virus (HIV) for any couple member;
* inseminations performed in a natural cycle or with clomiphene citrate (CC)

Ages: 20 Years to 44 Years | Sex: Female
Age Groups: Adult
Study Population: All couples attending our reproductive medical center to obtain homologous IUI program with COS between January 2007 and August 2014 ll couples had undergone a standard infertility evaluation, which included medical history, physical examination, and assessment of tubal patency by either hysterosalpingography or laparoscopy and hormonal analysis on cycle day 3.
Sampling Method: Probability Sample
Enrollment: 1251 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Success factors in the ovarian stimulation | 7 years
  The objective of this study is to evaluate the level of success factors of intrauterine insemination (IUI) in controlled ovarian stimulation (COS) in order to define the type of infertility. This retrospective cohort study included 1251 couples undergoing homologous IUIs.

CONTACTS AND LOCATIONS:
Overall Officials: Moncef Ben Khlifa, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No